CLINICAL TRIAL: NCT01274247
Title: Time of Cry After Lingual Frenotomy in Infants With Lingual Frenulum and Breastfeeding Difficulties, With or Without Use of Topical Benzocaine Analgesia
Brief Title: Use of Topical Benzocaine for Analgesia in Lingual Frenotomy of the Newborn
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study ethics committee recommended concluding the study for longer crying time with benzocaine and very short crying time in all participants.
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-SD-0385-CTIL
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Neonatal Tongue-tie; Maternal Nipple Pain Upon Breastfeeding; Neonatal Latch Difficulties
Keywords: Tongue-tie; Ankyloglossia
MeSH Terms: conditions — Ankyloglossia | interventions — Benzocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Benzocaine (Active Comparator): For infants treated with topical benzocaine prior to the procedure
  Interventions: Drug: Topical Benzocaine
- no benzocaine (No Intervention): No benzocaine applied

INTERVENTIONS:
Drug: Topical Benzocaine — Topical administration of a drop of benzocaine to the lingual frenulum
  Arms: Topical Benzocaine

SUMMARY:
Frenotomy of tongue-tie is commonly performed to resolve breastfeeding difficulties, eg maternal nipple pain and infant's latching difficulties. The procedure carries minor discomfort for the infants. It is not known whether the use of topical benzocaine, a very bitter tasting material' applied to the tongue-tie would decrease the length of cry. We will measure the duration of crying in infants treated with topical benzocaine to the duration in those not treated with the mediation.

ELIGIBILITY:
Inclusion Criteria:

* Full term Newborn infant
* Tongue-tie upon physical examination
* Maternal complains of nipple pain or difficult latch

Exclusion Criteria:

* Abnormal oral or nasopharyngeal anatomy
* Any known congenital malformations
* Prematurity

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Duration of cry after lingual frenotomy | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Dollberg, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Department of Neonatology, Tel AViv Medical Center, Tel Aviv, Israel